CLINICAL TRIAL: NCT01428960
Title: Acute Effects of Sn-1 and Sn-3 Palmitic Acid-rich or Stearic Acid-rich Fats on Postprandial Lipemia, Haemostatic and Inflammatory Markers, Gut Hormone Concentrations, Satiety, and Insulinemic Response in Human Volunteers
Brief Title: Study of Acute Effects of Sn-1 and Sn-3 Palmitic Acid-rich or Stearic Acid-rich Fats on Metabolic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: IMU University, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IMU R 069/2011
Record Dates: First submitted 2011-08-26; First posted 2011-09-05 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Palm mid fraction; Shea butter; sn-1, sn-3 fatty acids; Cholesterol; Postprandial lipemia,; Inflammatory markers; Satiety; Gut hormone; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Palm Mid Fraction (Experimental)
  Interventions: Dietary Supplement: Palm Mid Fraction, Shea Butter, High Oleic Sunflower Oil
- Shea Butter (Experimental)
  Interventions: Dietary Supplement: Palm Mid Fraction, Shea Butter, High Oleic Sunflower Oil
- High Oleic Sunflower Oil (Experimental)
  Interventions: Dietary Supplement: Palm Mid Fraction, Shea Butter, High Oleic Sunflower Oil

INTERVENTIONS:
Dietary Supplement: Palm Mid Fraction, Shea Butter, High Oleic Sunflower Oil — Acute effect of sn-1 and sn-3 palmitic acid-rich or stearic acid-rich fats on postprandial lipemia, haemostatic and inflammatory markers, gut hormone concentrations, satiety, and insulinemic response in human volunteers ; 6 wk each with 2 week wash out in between
  Other Names: POP vs SOS vs OOO

SUMMARY:
To determine the effect of degree of fat saturation on postprandial lipemia, haemostatic and inflammatory markers, gut hormone concentrations, satiety perceptions, and insulinemic responses in healthy adult subjects.

Study hypothesis: The degree of fat saturation does not affect postprandial lipemia, haemostatic and inflammatory markers, gut hormone concentrations, insulinemic or satiety responses in health adult subjects.

DETAILED DESCRIPTION:
The experimental are comprise of 50g fat, 14g protein and 84g carbohydrate. Each of the test fat [palm mid fraction (PMF), shea butter (SB) and high oleic sunflower oil (HOSF)] will be compared which will be in a form of experimental meals (muffin).

33 volunteers receives 3 experimental meals (muffins) in a random order, 2 week apart, over a 6-week period. They will be randomized, blinded and will undergo a 3x3 arms crossover. The first 15-ml ("0" min) fasting venous blood samples is obtained. Immediately thereafter, the subject consumes the test meal plus a glass of water within 15 minutes. The time sequence is started mid-way of consuming the test meal.

At 30 min, 60 min, 90, 120 min (2 hr), 150 min and 180 min (3 hr), 210 min, and 240 min (4 hr), 15-ml each of blood is collected (via a vascular catheter inserted earlier in the subjects hand/arm).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female staff, aged between 25-50 years
2. BMI 18.5 - 25.0 kg/m2
3. Blood pressure: Systolic: <140 mmHg, diastolic: <90 mmHg

c. Normolipidemic (Total cholesterol <6.2 mM/L (<240 mg/dL), Fasting TG <1.70 mM/L (<150 mg/dL) d. Fasting glucose 4.0- 7.0 mM/L

Exclusion Criteria:

1. Smokers
2. On cholesterol or blood glucose medication
3. Substance abuse (eg. alcohol, cigarette smoking)
4. For women, pregnant or lactating
5. Going overseas during period of study
6. Blood clotting problem
7. Public transportation to work

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
glucose-dependent insulintropic polypeptide (GIP) | 4 hours

SECONDARY OUTCOMES:
Lipid profile | 4 hours
Inflammatory markers | 4 hours
Haemostatic indices | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tony Ng, Principal Investigator — IMU University, Malaysia
Locations (1):
- Malaysian Palm Oil Board Kajang, Selangor,, Kajang, Selangor, Malaysia